CLINICAL TRIAL: NCT07054047
Title: Improving the Prognostic Accuracy of Staging Rectal Cancer Using Magnetic Resonance Imaging (MRI) - Detected Tumour Deposits and Vascular Invasion (mrTDV) Instead of Tumour Nodal Metastasis (mrTNM)
Brief Title: Improving Diagnosis and Treatment for Patients With Rectal Cancer
Acronym: MERCURY 3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: NHS England (Other Government); Pelican Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: EDGE: 176847; 348532 (Other: IRAS); 25/EM/0105 (Other: East Midlands - Derby Research Ethics Committee)
Record Dates: First submitted 2025-06-17; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: GI Cancer
Keywords: Shared decision making; Radiotherapy; Quality of Life; MRI Staging; MDT Decision Making; Histopathological Staging; Rectal Cancer; Preoperative staging
MeSH Terms: conditions — Gastrointestinal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will proceed through three phases: pre-intervention, intervention, and post-implementation.
  Pre-intervention - local MDT decisions based on current MRI reporting practices will be collected for six months.
  Intervention - local radiologists will be trained to recognize features of mrTDV and use a standardised reporting template. We will present the retrospective and radiologists' cohort results to MDT stakeholders who will agree the optimum stage based preoperative treatment decision making policy. We will offer training as required using the 2019 retrospective cohort.
  Post-intervention - local MDT decisions based on the consensus optimum stage based preoperative decision-making policy will be collected for six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm Schedule (No Intervention): All sites will begin in the Control arm, with patients recruited to the Control Arm Schedule. Clinical investigations prior to treatment, during treatment, after surgery and during further treatment should be performed as per standard clinical practice and as clinically indicated. Each site will remain in the Control Arm Schedule for six months. There will be a transition month with no recruitment where training is undertaken. After the transition month patients are recruited to the Intervention Arm Schedule . Patients will be recruited to either the Control or Intervention arms dependent on which arm is in progress at the site at the time of recruitment. There will be no crossover of patients between the arms at any point.
- Intervention Arm Schedule (Experimental): During the transition month, all Radiologists involved in reporting rectal cancers for the MDT will be offered training in reporting of mrTDV. Results of the retrospective data analysis will be shared at the MDT teams stakeholder meeting to determine their optimum stage based preoperative treatment decision making policy. Every site will remain in the Intervention Arm Schedule for six months.
  Patients will be recruited to either the Control or Intervention arms dependent on which arm is in progress at the site at the time of recruitment. There will be no crossover of patients between the arms at any point.
  Interventions: Other: mrTDV
- Retrospective cohort (No Intervention): Registration of all rectal cancer patients staged as non-metastatic in their site pre-treatment MDT from 1st January 2019 - 31st December 2019 should commence as soon as the site is issued the green light. The analysis of this data will be presented to their site MDT six months from the green light. Therefore, every effort should be made to complete the 2019 retrospective cohort registrations within the first three months of the trial start. We anticipate the average number of 2019 retrospective cohort patients treated for rectal cancer will be 20 per site.

INTERVENTIONS:
Other: mrTDV — The training of radiologists to implement specialised MRI reporting using the TDV staging system
  Arms: Intervention Arm Schedule

SUMMARY:
The cancer stage information from scans guides pre-operative treatment and the type of surgery offered. The investigators are studying whether a new Magnetic Resonance Imaging (MRI) staging method can improve the accuracy of prognosis for patients diagnosed with rectal cancer. The investigators will provide consultant radiologists with the know-how to report MRI scans using this new method and compare this with the existing method. This study will test this by comparing how accurately the old versus new method predict the outcomes of patients. The existing method relies on radiologists determining if tumour has spread through the bowel wall or not and whether there are suspected malignant lymph nodes. The new method looks for tumour spread into the veins and whether or not there are tumour deposits. Our previous research has shown that the new method is much more accurate at predicting prognosis, but this finding needs to be verified by a larger multicentre study.

The investigators are also studying the patient journey, so the investigators can better understand patients' experiences and the impact that treatments have on their quality of life. The investigators wish to understand if improvements in the accuracy of prognosis from scans could change treatment decisions in future. The investigators will also compare the radiology scan prediction of prognostic factors by looking carefully at the tumour specimens.

DETAILED DESCRIPTION:
A Retrospective and Prospective Cohort study to improve the prognostic accuracy of preoperative staging in patients diagnosed with primary rectal cancer. The intervention is the training of radiologists to implement specialised MRI reporting using the TDV staging system.

The investigators will collect anonymized scans, clinical and histopathology data from all rectal cancer patients diagnosed in 2019. The central reviewing radiologist will stage the scans by a) mrTDV and b) mrTNM into poor and good prognosis categories. The investigators will compare survival outcomes from original reports as well as the two staging systems using Kaplan-Meier and Cox Proportional-Hazard methods.

The investigators will compare prospectively collected data before and after implementation of the consensus for identifying and treating high-risk and low-risk rectal cancers. The investigators will report on the comparisons of staging, histopathology, MDT treatment decisions, resource utilisation, how patients experienced information provided for shared decision making before and after the intervention changes and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

1. Have a rectal cancer proven on biopsy or subsequent surgery
2. Sites able to submit anonymised MRI staging scans, pathology and imaging reports for central review
3. Aged 16 years or over

Exclusion Criteria:

1. Have irresectable metastatic disease at time of initial staging
2. Undergoing palliative treatment for Rectal Cancer
3. Have a biopsy-proven rectal malignancy which is not adenocarcinoma
4. Are contraindicated for MRI staging

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Validate that mrTDV staging can predict prognosis more accurately than mrTNM. | 1 and 5 years
  Survival differences for mrTNM and mrTDV before and after intervention will be compared

SECONDARY OUTCOMES:
Assess the degree of agreement between radiologists using mrTDV method of staging rectal cancer vs mrTNM method of staging rectal cancer. | 1 and 5 years
  Compare percentage agreement between radiologists when the TNM system of staging (scoring tumour, nodes and metastases) versus when using TDV system of staging (scoring tumour deposits and extramural venous invasion) is used.
Compare percentage agreement when staging of tumours using mrTDV method of staging rectal cancer and TNM method of staging rectal cancer with respective histopathology staging for prognosis. | 1 and 5 years
  Compare agreement in prognostic accuracy between radiology and histopathology using when the TNM system of staging (scoring tumour, nodes and metastases) versus when using TDV system of staging (scoring tumour deposits and extramural venous invasion) is used.
Measure the introduction of mrTDV staging and its impact on MDT decision-making with regards to treatment decisions | 1 and 5 years
  Comparison of what and how many treatments are offered as MDT policy to patients before and after mrTDV intervention
Report changes in numbers of treatments offered following MRI-TDV staging intervention | 6 months and 1 year
  Comparison of treatments given before and after mrTDV intervention
Report differences in disease free survival outcomes for rectal cancers staged using mrTNM method of staging versus TDV method of staging | 1 and 5 years
  Comparison of numbers of patients with disease free survival before and after mrTDV intervention
Report differences in local recurrence rates for rectal cancers staged using mrTNM method of staging versus TDV method of staging | 1 and 5 years
  Comparison of numbers of patients with local recurrencebefore and after mrTDV intervention
Qualitative EORTC QLQ-CR29 Questionnaire on Quality of Life of patients before and after adoption of mrTDV staging | 6 months, 1 and 5 years
  Comparison of QoL EORTC QLQ-CR29 scores before and after intervention. Questions relate to difficulty in performing every day tasks answers are rated 'Not at all' 'A Little' 'Quite a Bit' 'Very Much'
Qualitative EORTC QLQ-CR30 Questionnaire on Quality of Life of patients before and after adoption of mrTDV staging | 6 months, 1 and 5 years
  Comparison of QoL EORTC QLQ-CR30 scores before and after intervention. Questions relate to the presences of symptoms over the previous week answers are rated 'Not at all' 'A Little' 'Quite a Bit' 'Very Much'
Report differences in patient LARS scores before and after adoption of mrTDV staging | 6 months, 1 and 5 years
  Comparison of LARS scores before and after intervention. Questions relate to bowel function answers are rated 'Not at all' 'A Little' 'Quite a Bit' 'Very Much'
Report differences in patient shared decision making (SDM) before and after adoption of mrTDV staging | 6 months, 1 and 5 years
  Comparison of SM-Q9 scores before and after intervention. Answers are rated from 1 very poor to 7 excellent
Validate an educational programme for radiologists and MDTs to improve MRI reporting with TDV staging. | 6 months and 1 year
  Percentage agreement of radiologists prognostic accuracy using mrTNM method of staging versus mrTDV method of staging
Comparison of inpatient costs between patients before and after intervention | 18 and 36 months
  Comparison of relative percentage histopathological biomarkers screening panels between patients identified by the radiologist on the report before and after intervention
Comparison of total cost of outpatient visits between patients before and after intervention | 18 and 30 months
  Comparison of total cost of outpatient episodes based on individual pathways before and after intervention
Number of patients without disease and/or without stoma before and after intervention | 18 and 30 months
  DFS and stoma free survival in patients based on individual pathways before and after intervention
Assessment of novel and existing histopathological biomarkers to improve prognostic and predictive markers | 6, 12, 18 months and 3, 5 years
  Comparison of relative percentage histopathological biomarkers screening panels between patients identified by the radiologist on the report before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, MD, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - Southampton General Hospital, Southampton, Hampshire
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Salisbury District Hospital, Salisbury, Wiltshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris EJA, Finan PJ, Spencer K, Geh I, Crellin A, Quirke P, Thomas JD, Lawton S, Adams R, Sebag-Montefiore D. Wide Variation in the Use of Radiotherapy in the Management of Surgically Treated Rectal Cancer Across the English National Health Service. Clin Oncol (R Coll Radiol). 2016 Aug;28(8):522-531. doi: 10.1016/j.clon.2016.02.002. Epub 2016 Feb 28. PMID 26936609
- [Background] Wilkinson E. NICE withdraws quality standard on colorectal cancer treatment after "lack of consensus". Lancet Oncol. 2022 Mar;23(3):333. doi: 10.1016/S1470-2045(22)00084-5. Epub 2022 Feb 10. No abstract available. PMID 35151414
- [Background] Lord AC, D'Souza N, Shaw A, Rokan Z, Moran B, Abulafi M, Rasheed S, Chandramohan A, Corr A, Chau I, Brown G. MRI-Diagnosed Tumor Deposits and EMVI Status Have Superior Prognostic Accuracy to Current Clinical TNM Staging in Rectal Cancer. Ann Surg. 2022 Aug 1;276(2):334-344. doi: 10.1097/SLA.0000000000004499. Epub 2020 Sep 15. PMID 32941279
- [Background] Lord AC, Corr A, Chandramohan A, Hodges N, Pring E, Airo-Farulla C, Moran B, Jenkins JT, Di Fabio F, Brown G. Assessment of the 2020 NICE criteria for preoperative radiotherapy in patients with rectal cancer treated by surgery alone in comparison with proven MRI prognostic factors: a retrospective cohort study. Lancet Oncol. 2022 Jun;23(6):793-801. doi: 10.1016/S1470-2045(22)00214-5. Epub 2022 May 2. PMID 35512720